CLINICAL TRIAL: NCT05363943
Title: Double Plating (DP) Fixation vs Distal Femoral Replacement (DFR) in the Management of Distal Femoral Fractures in Geriatric Patients.
Brief Title: DP Vs DFR for Management of Geriatric Distal Femur Fractures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amr Gamaleldin Mahmoud Khalil Gendya (Other)
Responsible Party: Sponsor-Investigator, Amr Gamaleldin Mahmoud Khalil Gendya, Assistant Lecturer , Ain Shams University., Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD 291/2019
Record Dates: First submitted 2022-04-27; First posted 2022-05-06 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Distal Femur Fracture; Geriatrics
Keywords: Distal femoral fractures; Double plating; Distal femoral replacement; Geriatrics
MeSH Terms: conditions — Femoral Fractures, Distal

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fixation (Active Comparator): open reduction and internal fixation by using lateral and medial plates.
  Interventions: Procedure: double plating
- Replacement (Experimental): excision of the distal part of femur and replacement with distal femoral prosthesis
  Interventions: Procedure: Distal femoral replacement

INTERVENTIONS:
Procedure: double plating — open reduction and internal fixation by using lateral and medial plates.
  Arms: Fixation
Procedure: Distal femoral replacement — excision of the distal part of femur and replacement with distal femoral prosthesis
  Arms: Replacement

SUMMARY:
The aim of this study was to compare the functional and radiological outcomes of fixation by using double plating technique versus replacement using distal femur tumor prothesis as a primary management for the distal femoral fractures in geriatric patients. The hypothesis was that the distal femoral replacement will yield better functional outcome and earlier rehabilitation and return to pre-injury level of activity.

DETAILED DESCRIPTION:
Geriatric distal femoral fractures represent a major challenge for the orthopedic surgeons, to the present days still there is no definite algorithm or specific guidelines that can be used accurately in the management of these fractures. Unlike hip fractures however, there is no widely accepted treatment algorithm or standard of care.

The surgical treatment of distal femoral fractures depends on both patient and fracture characteristics. Options include conservative treatment, open reduction internal fixation, intramedullary nails, or recently distal femoral replacement.

There is currently a move towards distal femoral replacement (DFR) for these complex fractures which has the potential benefit of allowing early weight bearing, and therefore aiming to prevent complications associated with immobility and non-union.

Using distal femoral replacement had yield good results in small case series, as it allows immediate full weightbearing, eliminate the risk of nonunion and may provide greater satisfaction scores. However, DFR has its own risks, most notably deep infection, and loosening. While a DFR is more costly compared with fixation plates and nails, the initial increased cost may be outweighed by faster rehabilitation and return to the patient's usual place of residence.

In the study, the investigators are aiming to compare the functional and radiological outcomes of fixation by using double plating technique versus replacement as a primary management for the geriatric distal femoral fractures.

ELIGIBILITY:
Inclusion Criteria:

* AO 33 A3 and 33 C fractures
* Age group ≥ 60 years
* Closed fractures
* Neurovascular intact

Exclusion Criteria:

* Open fractures
* Non ambulant patients
* Patients with peripheral neurovascular diseases
* Peri-prosthetic fractures
* Associated other orthopedic injuries
* Poly-traumatized patients
* Pathological fractures

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
change in Knee Society Score | 1 month, 6 month and 12 month
  the score has two-part, knee and function parts. The score is graded from 0 to 100 in each domain with 100 is the best outcome and 0 is the worst. The knee part assesses the range of motion, pain, and alignment of the joint while the function part assesses walking, stairs and usage of walking aids.

SECONDARY OUTCOMES:
change in Knee range of motion | 1 month and 12 month
  Assessment of range of motion of the knee which has normal range from 0 to 135
Postoperative complications | form first day to 12 month
  Assessment of postoperative complications either early or late complications
Reoperation rate | form first day to 12 month
  Recording the need for secondary operation for a cause related to the fracture union, postoperative complications, or prothesis problems.
Operative time | At the operation
  Recording of the operative time from the time of incision to the time of skin closure

CONTACTS AND LOCATIONS:
Overall Officials: Amr GM Gendya, MSc Ortho., Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University - Faculty of Medicine, Cairo, Egypt